CLINICAL TRIAL: NCT05065385
Title: The EveryPrem Project: Evaluating the INTER-NDA for Standardized Neurodevelopmental Screening at 2 Years of Age for Children Born Preterm.
Acronym: EveryPrem
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Giancarlo Natalucci (Other)
Responsible Party: Sponsor-Investigator, Giancarlo Natalucci, Prof. Dr. med., University of Zurich
Organization: University of Zurich (Other)
Other Study IDs: BASEC 2020-02598
Record Dates: First submitted 2021-09-22; First posted 2021-10-04 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Prematurity
Keywords: Prematurity; Neurodevelopement; Follow-up; Screening; INTER-NDA
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: INTER-NDA — Neurodevelopmental Screening Test at age 2 years.
  Other Names: Bayley Scales of Infant and Toddler Development, 3rd Edition

SUMMARY:
Neurodevelopmental follow-up of infants at high-risk such as preterm born is necessary in order to early detect impairments and early start a supportive/therapeutic intervention. Valid tools should be available for screening infants with developmental problems even where resources are limited. Such screening would ensure an adequate medical care during and after hospital discharge as well as evidence-based parental pre- and postnatal counselling. While in Switzerland, these tools are specifically needed for the neurodevelopmental surveillance of moderate to late pretem born infants, in low- and mid-income countries, they are needed to monitor the whole population of preterm born infants.

To fill this important gap, the present study aims to determine whether it is feasible to extend neurodevelopmental screening (currently offered to only a very small part of children born preterm), by using a new cost-effective neurodevelopmental assessment, the INTERGROWTH-21st Neurodevelopment Assessment (INTER-NDA, www.inter-nda.com Assessment) at age 2 years.

DETAILED DESCRIPTION:
The pirmary objectives of the study are:

1. In very preterm born infants (born < 32 weeks' gestation)

   - To assess the concurrent validity of the INTER-NDA with the Bayley-III[13] at 2 years of corrected age in VPT infants.
2. In moderate to late preterm infants (born between 32 and 36 weeks' gestation) - To screen neurodevelopment performances at corrected 2 years of corrected age in MLPT infants by means of the INTER-NDA and to compare values with international INTER-NDA standard values.

ELIGIBILITY:
Inclusion Criteria:

* Former patient of the Department of Neonatology of the University Hospital Zurich
* Born between 01.01.2019 and 31.12.2021, i.e. aged 18 to 30 months at the time of the research visit
* Gestational age below 370/7 weeks
* Parent consent

Exclusion Criteria:

* Genetically defined syndrome (including chromosomal aberration) or inborn error of metabolism adversely influencing life expectancy or neurodevelopment.
* Major congenital malformations requiring surgical correction or potentially affecting neurodevelopmental outcome.
* Hypoxic ischemic encephalopathy after perinatal asphyxia defined as grade 2 or 3 according to Sarnat and Sarnat[19].
* Neonatal drug withdrawal syndrome or known maternal substance consumption of following illicit drugs during pregnancy: cocaine, heroin, Lysergic acid diethylamide (LSD), 3,4-Methylenedioxymethamphetamine (ecstasy), phencyclidine (PCP), and other amphetamine/methamphetamine.
* Children of parents who are not speaking German

Ages: 18 Months to 30 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All preterm born infants (i.e. born at < 37 weeks' gestation) who were either born at or received neonatal care at the University Hospital Zurich in 2019-2021 are eligible for the present study.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
INTER-NDA domain scores and centiles | At age 18 to 20 months; test duration 15 to 20 minutes.
  The INTERGROWTH-21st Neurodevelopment Assessment (INTER-NDA) is new cost-effective neurodevelopmental assessment for 2-year old infants.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF